CLINICAL TRIAL: NCT01763242
Title: EMAN-Anaemia: An Open Labelled Randomised Control Trial of the Synchronized Electronic MANagement of Anaemia in Chronic Kidney Disease (CKD) Compared to Usual Care Anaemia Management
Brief Title: Study of the Effect of Synchronised Anaemia Management in Chronic Kidney Disease
Acronym: EMAN-Anaemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Western Health, Australia (Other Government)
Responsible Party: Principal Investigator, Dr Craig Nelson, Head of Unit - Nephrology, Western Health, Australia
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HREC: 2010.267
Record Dates: First submitted 2013-01-06; First posted 2013-01-08 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Kidney Failure, Chronic; Anemia
Keywords: CKD, Anaemia, Synchronization, Monthly dosing, Home Delivery
MeSH Terms: conditions — Kidney Failure, Chronic; Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- EMAN (Active Comparator): Electronic auditing via synchronised blood tests and monthly dosing ESA and Home delivery of ESA from Pharmacy if required
  Interventions: Other: EMAN
- Control (No Intervention): Standard Outpatient Care with usual blood tests and follow up, and varied ESA dosing and frequency times. Patients are responsible for collecting their own ESA from Pharmacy

INTERVENTIONS:
Other: EMAN — See details on ESA Synchronization and Dosing in Detailed Description Above
  Other Names: Synchronised Blood Testing; Electronic upload of Blood Results; Synchronised ESA dosing monthly; Home delivery of ESA
  Arms: EMAN

SUMMARY:
Aims:

1. To establish an electronic process for CKD anaemia management using monthly synchronized dosing of erythrocyte stimulating agents (ESA).
2. To compare this electronic process with "present anaemia management" in the traditional outpatient setting.
3. To monitor Hb targets and clinical endpoints of study groups to model a larger multicentre study focusing on these endpoints.

DETAILED DESCRIPTION:
CKD Stages 3 to 5 Subjects will be randomised and stratified according to Age, Gender, CKD Stage, Known Cardiovascular Disease, Diabetes and ESA Type into EMAN vs. Control

Details of EMAN synchronization and Dosing:

Monthly dose of ESA is calculated by:

Monthly dose = present dose x (28/present frequency (days))

Synchronization will be achieved by using the formula: "Synchronization dose of ESA = (28-Days until next injection is due)/28 x monthly dose of ESA

The dose of ESA/C.E.R.A. should be adjusted to maintain the individual patient's haemoglobin within a range of 11± 1.0 g/dL of the reference haemoglobin concentration ie. between 10.0 and 12.0 g/dL

Haemoglobin Value Corrective Adjustment

* A single value >13 g/dL Interrupt treatment until Hb falls below 12 g/dL then re-start treatment at 50% of previous dose
* A single value <9 g/dL Increase dose by 50%
* Difference between two consecutive Hb values indicates ≥2 g/dL increase Reduce dose by 50%
* Difference between two consecutive Hb values indicates ≥2 g/dL decrease Increase dose by 50%
* >11.5 g/dL and <13 g/dL AND deviation from reference value is >1g/dL. Reduce dose by 25%
* <10.5 g/dL and >9 g/dL AND deviation from reference value is >1g/dL. Increase dose by 25%
* >12 g/dL Reduce dose by 25%
* <10 g/dL Increase dose by 25%

Statistics:

Audit of present practice suggests CKD patients achieve only 30% on target (Hb 10-12g/dL) while well audited dialysis units in our service can achieve 60% at target.

If an improvement from 30% to 60% is expected in the EMAN verses Control arm then 100 patients (50 in each group) would be required to show a significant difference p<0.05 with 85% power.

Patients will be analysed on an intention to treat basis Primary and Secondary Endpoint data will be compared between study and control groups using unpaired student t-tests after normalisation of data as required and/or chi squared analysis.

Statistical significance will be taken at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age > 18 years
* Chronic renal anaemia already on ESA therapy as defined by Pharmaceutical Benefits Scheme Criteria

Exclusion Criteria:

* Pregnancy
* Significant acute bleeding such as overt gastrointestinal bleeding
* A known haematological cause for anaemia
* Known metastatic malignancy
* Present participation in another interventional clinical trial • Known hypersensitivity to recombinant human erythropoietin, polyethylene glycol or to any constituent of the study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2011-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Haemoglobin | 12 months
  Haemoglobin (Hb) Targets: % above/within/below target ; % Time Hb above/within/below Target ie. Hb 10 to 12g/dL.

SECONDARY OUTCOMES:
All Cause Hospitalisation | 12 months
  Same day and Non Same Day Hospitalisation analysis, Total Hospitalisations
Outpatient Review Numbers | 12 months
Primary Care review Numbers | 12 months
Cardiovascular Hospitalisation | 12 months
Cerebrovascular Hospitalisation | 12 months
Peripheral Vascular Hospitalisation | 12 months
Thrombosis Events | 12 months
  Venous and Arterial
Renal Replacement Therapy Commencement | 12 months
  Dialysis and Renal transplantation
Deaths | 12 months
Quality of Life | 12 months
Missed Doses of ESA | 12 months
Fe Targets | 12 months
Blood Transfusion Numbers | 12 months
Fe Transfusion Numbers | 12 months
Total Adverse Events | 12 months
Anaemia Co-Ordinator Time | 12 months
Pharmacy Time | 12 months
Courier Costs | 12 months
Ambulance Transfer Numbers | 12 months
Cardiac and Vascular Biomarker Analysis | 12 months
  N Terminal Pro-Brain Natruretic Peptide, Interleukin-6, Tumour Necrosis Factor alpha, High Sensitivity C Reactive Protein

OTHER OUTCOMES:
Sub-Analysis of Outcomes by ESA Type | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Craig L Nelson, MBBSFRACPPhD, Principal Investigator — Western Health, Australia
Locations (1):
- Western Health, Footscray, Victoria, Australia